CLINICAL TRIAL: NCT04510623
Title: Host Response Mediators in Coronavirus (COVID-19) Infection - Is There a Protective Effect of Angiotensin II Type 1 Receptor Blockers (ARBs) on Outcomes of Coronavirus Infection?
Brief Title: Host Response Mediators in Coronavirus (COVID-19) Infection
Acronym: ARBS CORONA I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); British Columbia Centre for Disease Control (Other Government); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); University of Toronto (Other); University of Ottawa (Other); University of Calgary (Other); University of Alberta (Other); University of Victoria (Other); Wuhan University (Other); Peking Union Medical College (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jim Russell, Study-Wide Principal Investigator, University of British Columbia
Other Study IDs: H20-00600
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; SARS-CoV2
Keywords: ARBs; angiotensin II type 1 receptor blocker; ACEi; acute respiratory distress syndrome; COVID-19; coronavirus; Multisite; Canada; Observational; acute kidney injury; shock
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Coronavirus Infections; Acute Kidney Injury; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID-19 Patients on ARBs: This is an observational cohort study. Those who have COVID-19 in hospital and are on Angiotensin Receptor Blockers will be included in this cohort.
  Interventions: Other: ARBs and/or ACE inhibitors
- COVID-19 Patients on ACE inhibitors: This is an observational cohort study. Those who have COVID-19 in hospital and are on Angiotensin-Converting Enzyme inhibitors will be included in this cohort.
  Interventions: Other: ARBs and/or ACE inhibitors
- COVID-19 Patients on ARBs or ACE inhibitors: This is an observational cohort study. Those who have COVID-19 in hospital and are on ARBs or ACEi's will be included in this cohort.
  Interventions: Other: ARBs and/or ACE inhibitors
- COVID-19 Patients not on ARBs or ACE inhibitors: This is an observational cohort study. Those who have COVID-19 in hospital and are not on ARBs or ACEi's will be included in this cohort.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ARBs and/or ACE inhibitors — This is an observational study only.
  Groups: COVID-19 Patients on ACE inhibitors; COVID-19 Patients on ARBs; COVID-19 Patients on ARBs or ACE inhibitors
Other: Usual Care — This is an observational study only.
  Groups: COVID-19 Patients not on ARBs or ACE inhibitors

SUMMARY:
The coronavirus (COVID-19) pandemic continues to grow exponentially. Angiotensin II levels are increased in human influenza and are associated with influenza viral load, disease progression and mortality. Preliminary data shows angiotensin II receptor blockers (ARBs) limits lung injury in murine influenza H7N9, as well as viral titre and RNA. ARBs could limit viral titre and organ injury in COVID-19. We will therefore collect clinical chart data and test angiotensin II levels of patients who are admitted to ICU with COVID-19 to determine whether there is a correlation between taking ARBs and clinical outcomes in these patients.

Other blood biomarkers and clinical risk factors for COVID-19 have come to light in recent weeks. We include these in our observational analysis to help generate an understanding of COVID-19 presentation and blood biomarker characterization of disease.

DETAILED DESCRIPTION:
Purpose: To determine whether angiotensin II receptor blockers (ARBs) decrease severity or mortality in hospitalized COVID-19 infected adults.

Main Hypothesis: Modulation of ACE2 by ARBs decreases the need for hospitalization, severity (need for ventilation, vasopressors, extracorporeal membrane oxygenation or renal replacement therapy) or mortality of hospitalized COVID-19 infected adults.

Secondary Hypotheses:

* Plasma angiotensin I and II and other biomarker levels are associated with effectiveness of ARBs in hospitalized COVID-19 adults
* Modulation of ACE2 by angiotensin type I receptor blockers is associated with decreased rate of hospitalization for COVID-19
* In patients already on ARBs when they are hospitalized continuing ARBs is associated with decreased World Health Organization (WHO) COVID-19 ordinal outcome scale

Justification: The COVID-19 epidemic continues to grow exponentially affecting over 71,429 individuals with 1775 deaths (February 17, 2020), mostly in China but also in other countries. The population mortality rate is 2% (lower than SARS (10%) and MERS (36%) but is 10% in hospitalized and 24% in ICU-admitted COVID-19 patients in China. Recent data from China (not yet public domain) suggest ICU mortality is higher (J. Marshall personal communication). Interventions to date include quarantine, isolation and usual clinical care. There are no proven antiviral or host modulating interventions for COVID-19. Notably, critically ill COVID-19 patients have similar mortality rates as sepsis and acute respiratory distress syndrome. Cohort studies have shown that patients already on angiotensin-converting enzyme (ACE) inhibitors and angiotensin II receptor blockers (ARBs) have lower sepsis mortality. Angiotensin II worsens lung injury in influenza models because ACE2 is downregulated in H1N1, H5N1, H7N9, and SARS viral infections leading to increased angiotensin II. Angiotensin II levels are increased in human influenza and are associated with influenza viral load, disease progression and mortality. Preliminary data shows ARBs limits lung injury in murine influenza H7N9, as well as viral titre and RNA. ARBs could limit viral titre and organ injury in COVID-19.

Research Design:

Prospective clinical chart review: we will collect clinical data on the participant throughout their hospital stay. Includes collection of baseline characteristics such as age, sex, heart rate, respiratory rate, temperature, blood pressure, SaO2, respiratory (PaO2/FiO2), renal (creatinine) and hepatic (bilirubin) function, use of oxygen, vasopressors, ventilation and RRT. They will be followed daily throughout their hospital stay, until death or discharge. Using left over clinical blood collected upon admission to hospital, plasma angiotensin I and II and other biomarker levels will be measured in our research laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age who have confirmed COVID-19 infection (according to local hospital or provincial laboratories clinically approved laboratory testing for COVID-19).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients with confirmed COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 WHO ordinal scale | 14 days

SECONDARY OUTCOMES:
Organ Dysfunction | 14 days
28-day mortality | 29 days or less (may be discharged from critical care before day 28)
Hospital/ICU length of stay | 29 days or less (may be discharged before day 28)
ICU admission | 29 days or less (may be discharged from critical care before day 28)

CONTACTS AND LOCATIONS:
Overall Officials: James A Russell, MD, Principal Investigator — St Paul's Hospital, Center for Heart and Lung Innovation
Locations (15):
- Canada (15):
  - University of Calgary - Foothills, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St Pauls Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
  - Queens University, Kingston, Ontario
  - Humber River Hospital, North York, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Lee T, Cheng MP, Vinh DC, Lee TC, Tran KC, Winston BW, Sweet D, Boyd JH, Walley KR, Haljan G, McGeer A, Lamontagne F, Fowler R, Maslove D, Singer J, Patrick DM, Marshall JC, Burns KD, Murthy S, Mann PK, Hernandez G, Donohoe K, Rocheleau G, Russell JA; ARBs CORONA I study investigators. Organ dysfunction and death in patients admitted to hospital with COVID-19 in pandemic waves 1 to 3 in British Columbia, Ontario and Quebec, Canada: a cohort study. CMAJ Open. 2022 Apr 19;10(2):E379-E389. doi: 10.9778/cmajo.20210216. Print 2022 Apr-Jun. PMID 35440485
- [Derived] Russell JA, Marshall JC, Slutsky A, Murthy S, Sweet D, Lee T, Singer J, Patrick DM, Du B, Peng Z, Cheng M, Burns KD, Harhay MO. Study protocol for a multicentre, prospective cohort study of the association of angiotensin II type 1 receptor blockers on outcomes of coronavirus infection. BMJ Open. 2020 Dec 7;10(12):e040768. doi: 10.1136/bmjopen-2020-040768. PMID 33293316